CLINICAL TRIAL: NCT01654016
Title: Study of Antiinflammatory Effects of Detralex (Daflon) in Patients With Chronic Venous Disease
Brief Title: Study of Antiinflammatory Effects of Detralex (Daflon)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Marko Ajduk, MD PhD, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Detra-001-Ajd
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Chronic Venous Insufficiency
Keywords: varicose veins; inflammation
MeSH Terms: conditions — Varicose Veins; Inflammation | interventions — S 5682; Diosmin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Detralex (Active Comparator): Detralex 500 mg twice daily for three month prior to surgery
  Interventions: Drug: Detralex
- Not taking Detralex (No Intervention): Not taking Detralex for three months prior to surgery

INTERVENTIONS:
Drug: Detralex — Detralex 500 mg twice daily for three month prior to surgery
  Other Names: Daflon
  Arms: Detralex

SUMMARY:
Aim of the study:

To investigate if there is a differences in expression of inflammatory markers in venous wall and blood among patients treated with Detralex and those not treated with Detralex (control group).

DETAILED DESCRIPTION:
Chronic venous disease (CVD) represents one of the most common vascular disorder. It's different clinical manifestations (most often seen as varicose veins) can be observed in up to 40% of adult female population and in about 30% of adult males.

Different mechanical and biological factors play role in the process of deterioration of venous wall tone and consequent vein valve disfunction that eventually lead to increase venous pressure . Evidence suggest that inflammation has a central place in this process even from the early stage of CVD.

Usual symptoms of venous insufficiency are pain, leg heaviness, night cramping, itching, and are often accompanied with leg edema. The extent of clinical manifestation may not correlate with patients' symptoms. Treatment of varicose veins encompasses vein surgery (stripping, phlebectomy, radiofrequency and laser ablation), sclerotherapy and compression therapy. Detralex (in some countries registered as Daflon) is an oral flavonoid that consists of 90% micronized diosmin and 10% flavonoids expressed as hesperidin. Several studies showed some beneficial effects of Detralex in alleviating symptoms in patients with CVD. It may be used in conjunction with surgery, sclerotherapy, or compression therapy or it may be the only therapy when other therapeutical modalities are not indicated or not feasable.

Animal studies showed antiinflammatory effects of Daflon in way that Daflon acts favorably on microcirculatory complications by normalizing the synthesis of prostaglandins and free radicals. It decreases bradykinin-induced microvascular leakage and inhibits leukocyte activation, trapping, and migration.

However, by searching the available literature (MEDLINE) we found no study that investigated what are the antiinflammatory effects of flavonoids in humans.

The aim of this study is to investigate if there is a differences in expression of inflammatory markers in venous wall and blood between patients treated with Detralex and those not treated with Detralex (control group).

ELIGIBILITY:
Inclusion Criteria:

* Chronic venous disease (CEAP 2 and 3) and saphenofemoral insufficiency

Exclusion Criteria:

* Previous deep venous thrombosis
* Previous or acute thrombophlebitis of the GSV (confirmed by duplex findings - morphologic changes of the GSV above the knee)
* Immunological disorders
* Diabetes type I or II,
* Severe inflammatory disease: such as Behcet, lupus, Horton and other arteritis, polyarthritis, spondylarthritis or sclerodermia
* Recent (less than 3 months) or scheduled non-authorized non-pharmacological treatments:
* Sclerotherapy,
* Surgical treatment of varicose veins (crossectomy, phlebectomy),
* Endovenous treatment (endovenous laser, radiofrequency),
* Non-authorized pharmacological treatment in the last 3 months and during the study:
* Anti-inflammatory agents (except acetylsalicylic acid at dose 350 mg daily),
* Systemic corticosteroids or immunosuppressives,
* Venoactive drugs including open label MPFF,
* Pentoxifylline
* Patients already (at the time of randomization) taking Detralex for symptoms linked to chronic venous disease
* Arterial insufficiency (absent pedal pulses or ABI < 0.9)
* Any important clinical or laboratory abnormalities
* Pregnancy, breastfeeding or wish of becoming pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-08; Primary Completion 2019-05 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Antiinflammatory Effects of Detralex (Daflon) | 14 months
  The following markers of inflammation will be analyzed:
  Blood (biochemical analysis): soluble ICAM-1, soluble VCAM-1, E-selectin, L selectin PAI-1, TIMP-1, Angiopoietin-1, Angiopoietin-2 and Tie-2.
  Vein wall ([immuno]histological and biochemical analysis) : CD 45 (leukocytes), S100 (C-fibers), MMP3, MMP9, SMC (smooth muscle cells). Presence (or not) of microthrombi in the vein lumen

SECONDARY OUTCOMES:
Clinical effects of Detralex (Daflon) | 14 months
  Subjective perception of pain, leg heaviness, cramping and itching will be assessed using visual analogue scale (VAS) graded from 0 to 10. Leg edema will be assessed by measuring the leg circumference. Data will be recorded as follow:
  1. three months before the surgery
  2. one day before the surgery
  3. one week after the surgery
  4. one month after bthe surgery
  5. three months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marko Ajduk, PhD, Principal Investigator — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] Eberhardt RT, Raffetto JD. Chronic venous insufficiency. Circulation. 2005 May 10;111(18):2398-409. doi: 10.1161/01.CIR.0000164199.72440.08. No abstract available. PMID 15883226
- [Background] Nicolaides AN. From symptoms to leg edema: efficacy of Daflon 500 mg. Angiology. 2003 Jul-Aug;54 Suppl 1:S33-44. doi: 10.1177/0003319703054001S05. PMID 12934755
- [Background] Sezer A, Usta U, Kocak Z, Yagci MA. The effect of a flavonoid fractions diosmin + hesperidin on radiation-induced acute proctitis in a rat model. J Cancer Res Ther. 2011 Apr-Jun;7(2):152-6. doi: 10.4103/0973-1482.82927. PMID 21768702
- [Background] Perrin M, Ramelet AA. Pharmacological treatment of primary chronic venous disease: rationale, results and unanswered questions. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):117-25. doi: 10.1016/j.ejvs.2010.09.025. Epub 2010 Dec 3. PMID 21126890
- [Background] Bergan JJ. Chronic venous insufficiency and the therapeutic effects of Daflon 500 mg. Angiology. 2005 Sep-Oct;56 Suppl 1:S21-4. doi: 10.1177/00033197050560i104. PMID 16193222
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449